CLINICAL TRIAL: NCT06171204
Title: Gebruik Van Stromale Vasculaire Fractie Uit Vetweefsel Na Invriezing Voor Knie Arthrose
Brief Title: The Use of Stromal Vascular Fraction for Knee Arthrosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-07772
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Knee Arthrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Injection of SVF in fat pad of the knee — Knee fat pad injection with SVF at orthopaedics/physical medicine outpatient clinic

SUMMARY:
A trial to investigate the safety and efficacy of SVF for the treatment of knee arthrosis.

Patients will undergo a single liposuction to obtain the SVF. The SVF will then be isolated and frozen in our laboratory. The SVF will then be injected up to 2 times into the fat pad of the patient's knee.

DETAILED DESCRIPTION:
Stromal Vascular Fraction (SVF) from adipose tissue is increasingly being used in the clinic for a variety of conditions (skin disorders, joint pain, etc.). SVF is a collective term for cells that can be obtained from liposuction fat. These cells can be separated from the fat by mechanical processing of the liposuction fat combined with an additional centrifugation.

Despite the fact that enough SVF can be isolated after such a liposuction for multiple treatments (>3), our research group has found a way to safely freeze SVF without significant loss of SVF cells. In this way, a patient would only have to undergo one liposuction and associated anesthesia to be able to obtain multiple SVF treatments.

ELIGIBILITY:
Inclusion Criteria:

* Legal capacity
* Osteochondral lesions
* Inflammatory complaints
* (Peri)tendinitis or tendinopathies and ligamentous injuries
* Impingement complaints
* Arthrofibrosis
* Anterior knee pain

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the safety of SVF injections after cryo preservation | 1 year
  The patient will complete the KOOS questionnaire (Knee Injury and Osteoarthritis Outcome Score) on several timepoints.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ GENT, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No